CLINICAL TRIAL: NCT01507831
Title: Long-term Safety and Tolerability of SAR236553 (REGN727) in High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Lipid Modifying Therapy: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Long-term Safety and Tolerability of Alirocumab (SAR236553/REGN727) Versus Placebo on Top of Lipid-Modifying Therapy in High Cardiovascular Risk Patients With Hypercholesterolemia (ODYSSEY Long Term)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTS11717; 2011-002806-59 (EudraCT Number); U1111-1121-3928 (Other: UTN)
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for alirocumab) every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for 78 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Lipid-Modifying Therapy (LMT)
- Alirocumab (Experimental): Alirocumab 150 mg Q2W added to stable LMT for 78 weeks.
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Placebo (for alirocumab) — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a pre-filled syringe.
  Arms: Placebo
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a pre-filled syringe.
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab
Drug: Lipid-Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9).

Primary Objective of the study:

To evaluate the long-term safety and tolerability of alirocumab in high cardiovascular risk participants with hypercholesterolemia not adequately controlled with their current lipid modifying therapy (LMT).

Secondary Objectives:

* To evaluate the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels after 24 weeks of treatment in comparison with placebo.
* To evaluate the effect of alirocumab in comparison with placebo on LDL-C at other time points.
* To evaluate the effects of alirocumab on other lipid parameters.

DETAILED DESCRIPTION:
The maximum study duration was to be 89 weeks per participant, including a 3-week screening period, a 78-week randomized treatment period and 8-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

Either A or B below and who were not adequately controlled with their lipid-modifying therapy:

A) Participants with heterozygous familial hypercholesterolemia (heFH) with or without established coronary heart disease (CHD) or CHD risk equivalents

OR

B) Participants with hypercholesterolemia together with established CHD or CHD risk equivalents.

Exclusion criteria:

* Age < 18 years
* LDL-C <70 mg/dL (< 1.81 mmol/L)
* Fasting serum triglycerides > 400 mg/dL (>4.52 mmol/L)

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2341 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (320):
- United States (115):
  - Investigational Site Number 840159, Huntsville, Alabama
  - Investigational Site Number 840028, Gilbert, Arizona
  - Investigational Site Number 840035, Sierra Vista, Arizona
  - Investigational Site Number 840052, Tempe, Arizona
  - Investigational Site Number 840065, Tempe, Arizona
  - Investigational Site Number 840079, Tempe, Arizona
  - Investigational Site Number 840094, Tempe, Arizona
  - Investigational Site Number 840103, Tucson, Arizona
  - Investigational Site Number 840209, Beverly Hills, California
  - Investigational Site Number 840194, Beverly Hills, California
  - Investigational Site Number 840207, Fresno, California
  - Investigational Site Number 840101, Lincoln, California
  - Investigational Site Number 840076, Long Beach, California
  - Investigational Site Number 840214, Pasadena, California
  - Investigational Site Number 840045, Sacramento, California
  - Investigational Site Number 840163, Santa Rosa, California
  - Investigational Site Number 840086, Colorado Springs, Colorado
  - Investigational Site Number 840077, Golden, Colorado
  - Investigational Site Number 840224, Bridgeport, Connecticut
  - Investigational Site Number 840134, Guilford, Connecticut
  - Investigational Site Number 840246, Hartford, Connecticut
  - Investigational Site Number 840055, Stamford, Connecticut
  - Investigational Site Number 840091, Stamford, Connecticut
  - Investigational Site Number 840150, Atlantis, Florida
  - Investigational Site Number 840020, Bradenton, Florida
  - Investigational Site Number 840041, Brandon, Florida
  - Investigational Site Number 840184, Clearwater, Florida
  - Investigational Site Number 840242, Clearwater, Florida
  - Investigational Site Number 840039, Clearwater, Florida
  - Investigational Site Number 840182, Crystal River, Florida
  - Investigational Site Number 840002, Daytona Beach, Florida
  - Investigational Site Number 840166, Daytona Beach, Florida
  - Investigational Site Number 840167, Fleming Island, Florida
  - Investigational Site Number 840090, Fort Lauderdale, Florida
  - Investigational Site Number 840018, Fort Lauderdale, Florida
  - Investigational Site Number 840153, Jacksonville, Florida
  - Investigational Site Number 840181, Jacksonville, Florida
  - Investigational Site Number 840152, Jacksonville, Florida
  - Investigational Site Number 840154, Lake Mary, Florida
  - Investigational Site Number 840059, Largo, Florida
  - Investigational Site Number 840221, Miami, Florida
  - Investigational Site Number 840021, New Port Richey, Florida
  - Investigational Site Number 840122, New Smyrna Beach, Florida
  - Investigational Site Number 840151, Ocala, Florida
  - Investigational Site Number 840108, Ormond Beach, Florida
  - Investigational Site Number 840067, Palm Harbor, Florida
  - Investigational Site Number 840006, Pembroke Pines, Florida
  - Investigational Site Number 840168, Ponte Vedra, Florida
  - Investigational Site Number 840164, Sarasota, Florida
  - Investigational Site Number 840175, Sarasota, Florida
  - Investigational Site Number 840001, St. Petersburg, Florida
  - Investigational Site Number 840003, St. Petersburg, Florida
  - Investigational Site Number 840036, West Palm Beach, Florida
  - Investigational Site Number 840117, Cumming, Georgia
  - Investigational Site Number 840110, Roswell, Georgia
  - Investigational Site Number 840026, Savannah, Georgia
  - Investigational Site Number 840075, Meridian, Idaho
  - Investigational Site Number 840027, Evansville, Indiana
  - Investigational Site Number 840093, Indianapolis, Indiana
  - Investigational Site Number 840222, Iowa City, Iowa
  - Investigational Site Number 840165, West Des Moines, Iowa
  - Investigational Site Number 840200, Kansas City, Kansas
  - Investigational Site Number 840040, Wichita, Kansas
  - Investigational Site Number 840061, Wichita, Kansas
  - Investigational Site Number 840032, Wichita, Kansas
  - Investigational Site Number 840084, Wichita, Kansas
  - Investigational Site Number 840244, Biddeford, Maine
  - Investigational Site Number 840158, Framingham, Maine
  - Investigational Site Number 840193, Novi, Michigan
  - Investigational Site Number 840162, Saginaw, Michigan
  - Investigational Site Number 840033, St Louis, Missouri
  - Investigational Site Number 840113, St Louis, Missouri
  - Investigational Site Number 840095, Henderson, Nevada
  - Investigational Site Number 840096, Henderson, Nevada
  - Investigational Site Number 840022, Edison, New Jersey
  - Investigational Site Number 840011, Hillsborough, New Jersey
  - Investigational Site Number 840049, Trenton, New Jersey
  - Investigational Site Number 840097, Bronxville, New York
  - Investigational Site Number 840129, Brooklyn, New York
  - Investigational Site Number 840160, Poughkeepsie, New York
  - Investigational Site Number 840217, Asheville, North Carolina
  - Investigational Site Number 840023, Charlotte, North Carolina
  - Investigational Site Number 840083, Greensboro, North Carolina
  - Investigational Site Number 840104, Raleigh, North Carolina
  - Investigational Site Number 840068, Cincinnati, Ohio
  - Investigational Site Number 840007, Dayton, Ohio
  - Investigational Site Number 840013, Marion, Ohio
  - Investigational Site Number 840161, Mentor, Ohio
  - Investigational Site Number 840005, Tulsa, Oklahoma
  - Investigational Site Number 840170, Beaver, Pennsylvania
  - Investigational Site Number 840180, Camp Hill, Pennsylvania
  - Investigational Site Number 840004, Duncansville, Pennsylvania
  - Investigational Site Number 840046, Jersey Shore, Pennsylvania
  - Investigational Site Number 840155, Phoenixville, Pennsylvania
  - Investigational Site Number 840177, Scranton, Pennsylvania
  - Investigational Site Number 840202, Wyomissing, Pennsylvania
  - Investigational Site Number 840073, Charleston, South Carolina
  - Investigational Site Number 840087, Greenville, South Carolina
  - Investigational Site Number 840074, Simpsonville, South Carolina
  - Investigational Site Number 840105, Varnville, South Carolina
  - Investigational Site Number 840190, Knoxville, Tennessee
  - Investigational Site Number 840092, Dallas, Texas
  - Investigational Site Number 840212, Dallas, Texas
  - Investigational Site Number 840058, Fort Worth, Texas
  - Investigational Site Number 840149, Fort Worth, Texas
  - Investigational Site Number 840070, Fort Worth, Texas
  - Investigational Site Number 840038, Houston, Texas
  - Investigational Site Number 840047, Houston, Texas
  - Investigational Site Number 840053, Plano, Texas
  - Investigational Site Number 840072, Sugar Land, Texas
  - Investigational Site Number 840241, Tyler, Texas
  - Investigational Site Number 840031, Salt Lake City, Utah
  - Investigational Site Number 840204, Chesapeake, Virginia
  - Investigational Site Number 840120, Spokane, Washington
  - Investigational Site Number 840111, Milwaukee, Wisconsin
- Argentina (6):
  - Investigational Site Number 032006, Buenos Aires
  - Investigational Site Number 032010, Caba
  - Investigational Site Number 032008, Capital Federal
  - Investigational Site Number 032001, Coronel Suárez
  - Investigational Site Number 032004, Resistencia
  - Investigational Site Number 032007, Zárate
- Belgium (4):
  - Investigational Site Number 056005, Antwerp
  - Investigational Site Number 056004, Genk
  - Investigational Site Number 056001, Natoye
  - Investigational Site Number 056002, Wetteren
- Bulgaria (9):
  - Investigational Site Number 100008, Pleven
  - Investigational Site Number 100014, Plovdiv
  - Investigational Site Number 100005, Sofia
  - Investigational Site Number 100012, Sofia
  - Investigational Site Number 100015, Sofia
  - Investigational Site Number 100009, Sofia
  - Investigational Site Number 100001, Sofia
  - Investigational Site Number 100013, Stara Zagora
  - Investigational Site Number 100007, Varna
- Canada (14):
  - Investigational Site Number 124013, Cambridge
  - Investigational Site Number 124027, Coquitlam
  - Investigational Site Number 124001, Hawkesbury
  - Investigational Site Number 124002, London
  - Investigational Site Number 124009, Mirabel
  - Investigational Site Number 124018, Montreal
  - Investigational Site Number 124007, Ottawa
  - Investigational Site Number 124011, Québec
  - Investigational Site Number 124008, Sarnia
  - Investigational Site Number 124005, St. John's
  - Investigational Site Number 124022, Terrebonne
  - Investigational Site Number 124003, Vancouver
  - Investigational Site Number 124006, Victoria
  - Investigational Site Number 124015, Woodstock
- Chile (4):
  - Investigational Site Number 152007, Osorno
  - Investigational Site Number 152008, Santiago
  - Investigational Site Number 152006, Santiago
  - Investigational Site Number 152004, Temuco
- Colombia (5):
  - Investigational Site Number 170004, Barranquilla
  - Investigational Site Number 170005, Barranquilla
  - Investigational Site Number 170008, Barranquilla
  - Investigational Site Number 170001, Manizales
  - Investigational Site Number 170003, Medellín
- Czechia (3):
  - Investigational Site Number 203004, Prague
  - Investigational Site Number 203007, Prague
  - Investigational Site Number 203006, Prague
- Denmark (5):
  - Investigational Site Number 208005, Aarhus
  - Investigational Site Number 208004, Hellerup
  - Investigational Site Number 208003, Slagelse
  - Investigational Site Number 208001, Svendborg
  - Investigational Site Number 208002, Viborg
- Finland (4):
  - Investigational Site Number 246002, Joensuu
  - Investigational Site Number 246001, Kokkola
  - Investigational Site Number 246003, Kuopio
  - Investigational Site Number 246004, Vantaa
- France (12):
  - Investigational Site Number 250007, Bandol
  - Investigational Site Number 250003, Broglie
  - Investigational Site Number 250014, Bron
  - Investigational Site Number 250004, Dijon
  - Investigational Site Number 250006, Lille
  - Investigational Site Number 250009, Nantes
  - Investigational Site Number 250001, Nantes
  - Investigational Site Number 250002, Paris
  - Investigational Site Number 250010, Pessac
  - Investigational Site Number 250012, Rennes
  - Investigational Site Number 250005, Vieux-Condé
  - Investigational Site Number 250008, Vihiers
- Germany (15):
  - Investigational Site Number 276001, Bad Wörishofen
  - Investigational Site Number 276007, Berlin
  - Investigational Site Number 276005, Berlin
  - Investigational Site Number 276014, Berlin
  - Investigational Site Number 276008, Bochum
  - Investigational Site Number 276009, Dresden
  - Investigational Site Number 276004, Essen
  - Investigational Site Number 276010, Frankfurt A.M.
  - Investigational Site Number 276011, Görlitz
  - Investigational Site Number 276019, Hanover
  - Investigational Site Number 276013, Leipzig
  - Investigational Site Number 276012, Magdeburg
  - Investigational Site Number 276003, Magdeburg
  - Investigational Site Number 276006, Schwerin
  - Investigational Site Number 276015, Witten
- Hungary (10):
  - Investigational Site Number 348003, Baja
  - Investigational Site Number 348007, Budapest
  - Investigational Site Number 348009, Budapest
  - Investigational Site Number 348008, Budapest
  - Investigational Site Number 348013, Budapest
  - Investigational Site Number 348004, Debrecen
  - Investigational Site Number 348002, Nagykanizsa
  - Investigational Site Number 348006, Nyíregyháza
  - Investigational Site Number 348001, Sopron
  - Investigational Site Number 348011, Úrhida
- Israel (4):
  - Investigational Site Number 376002, Afula
  - Investigational Site Number 376003, Holon
  - Investigational Site Number 376005, Holon
  - Investigational Site Number 376004, Nazareth
- Italy (8):
  - Investigational Site Number 380006, Chieti
  - Investigational Site Number 380002, Cinisello Balsamo
  - Investigational Site Number 380009, Milan
  - Investigational Site Number 380007, Napoli
  - Investigational Site Number 380001, Palermo
  - Investigational Site Number 380005, Pozzilli
  - Investigational Site Number 380008, Vittorio Veneto
  - Investigational Site Number 380010, Zingonia-Osio Sotto
- Mexico (7):
  - Investigational Site Number 484010, Df
  - Investigational Site Number 484004, México
  - Investigational Site Number 484008, Not Provided
  - Investigational Site Number 484001, San Luis Potosí City
  - Investigational Site Number 484002, Tijuana
  - Investigational Site Number 484009, Torreón
  - Investigational Site Number 484003, Xalapa
- Netherlands (12):
  - Investigational Site Number 528013, Amsterdam
  - Investigational Site Number 528001, Amsterdam
  - Investigational Site Number 528004, Breda
  - Investigational Site Number 528005, Eindhoven
  - Investigational Site Number 528007, Groningen
  - Investigational Site Number 528011, Hoogeveen
  - Investigational Site Number 528002, Hoorn
  - Investigational Site Number 528008, Leiderdorp
  - Investigational Site Number 528009, Rotterdam
  - Investigational Site Number 528006, Velp
  - Investigational Site Number 528012, Venlo
  - Investigational Site Number 528010, Zoetermeer
- Norway (5):
  - Investigational Site Number 578005, Elverum
  - Investigational Site Number 578001, Hamar
  - Investigational Site Number 578002, Oslo
  - Investigational Site Number 578004, Skedsmokorset
  - Investigational Site Number 578003, Stavanger
- Poland (9):
  - Investigational Site Number 616008, Gdynia
  - Investigational Site Number 616003, Gdynia
  - Investigational Site Number 616001, Gniewkowo
  - Investigational Site Number 616010, Katowice
  - Investigational Site Number 616018, Krakow
  - Investigational Site Number 616004, Piotrkow Trybunalski
  - Investigational Site Number 616013, Puławy
  - Investigational Site Number 616009, Warsaw
  - Investigational Site Number 616007, Wroclaw
- Portugal (4):
  - Investigational Site Number 620006, Funchal / Madeira
  - Investigational Site Number 620002, Lisbon
  - Investigational Site Number 620001, Lisbon
  - Investigational Site Number 620005, Porto
- Romania (4):
  - Investigational Site Number 642005, Baia Mare
  - Investigational Site Number 642002, Brasov
  - Investigational Site Number 642004, Târgu Mureş
  - Investigational Site Number 642001, Timișoara
- Russia (7):
  - Investigational Site Number 643005, Barnaul
  - Investigational Site Number 643012, Moscow
  - Investigational Site Number 643008, Moscow
  - Investigational Site Number 643014, Perm
  - Investigational Site Number 643006, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643004, Yaroslavl
- South Africa (11):
  - Investigational Site Number 710010, Centurion
  - Investigational Site Number 710008, Meyerspark
  - Investigational Site Number 710011, Middelburg
  - Investigational Site Number 710006, Parktown
  - Investigational Site Number 710004, Pretoria
  - Investigational Site Number 710001, Pretoria
  - Investigational Site Number 710002, Pretoria
  - Investigational Site Number 710009, Roodepoort
  - Investigational Site Number 710003, Somerset West
  - Investigational Site Number 710005, Witbank
  - Investigational Site Number 710007, Worcester
- Spain (8):
  - Investigational Site Number 724006, Córdoba
  - Investigational Site Number 724003, Granada
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724007, Málaga
  - Investigational Site Number 724008, Quart de Poblet
  - Investigational Site Number 724005, Reus
  - Investigational Site Number 724001, Sabadell
  - Investigational Site Number 724004, Seville
- Sweden (5):
  - Investigational Site Number 752001, Örebro
  - Investigational Site Number 752002, Rättvik
  - Investigational Site Number 752006, Stockholm
  - Investigational Site Number 752003, Stockholm
  - Investigational Site Number 752004, Stockholm
- Ukraine (11):
  - Investigational Site Number 804012, Chernivtsi
  - Investigational Site Number 804003, Dnipropetrovsk
  - Investigational Site Number 804002, Donetsk
  - Investigational Site Number 804014, Kharkiv
  - Investigational Site Number 804016, Kiev
  - Investigational Site Number 804011, Kyiv
  - Investigational Site Number 804010, Kyiv
  - Investigational Site Number 804001, Kyiv
  - Investigational Site Number 804008, Kyiv
  - Investigational Site Number 804013, Kyiv
  - Investigational Site Number 804005, Zhytomyr
- United Kingdom (19):
  - Investigational Site Number 826004, Addlestone
  - Investigational Site Number 826009, Birmingham
  - Investigational Site Number 826016, Birmingham
  - Investigational Site Number 826021, Blackpool
  - Investigational Site Number 826023, Cambridge
  - Investigational Site Number 826012, Cardiff
  - Investigational Site Number 826024, Chichester
  - Investigational Site Number 826006, Chorley
  - Investigational Site Number 826010, Glasgow
  - Investigational Site Number 826003, Irvine
  - Investigational Site Number 826008, Liverpool
  - Investigational Site Number 826005, Liverpool
  - Investigational Site Number 826025, Manchester
  - Investigational Site Number 826007, Manchester
  - Investigational Site Number 826001, Middlesex
  - Investigational Site Number 826019, Penzance
  - Investigational Site Number 826011, Reading
  - Investigational Site Number 826013, Romford
  - Investigational Site Number 826014, Soham

REFERENCES:
- [Result] Robinson JG, Farnier M, Krempf M, Bergeron J, Luc G, Averna M, Stroes ES, Langslet G, Raal FJ, El Shahawy M, Koren MJ, Lepor NE, Lorenzato C, Pordy R, Chaudhari U, Kastelein JJ; ODYSSEY LONG TERM Investigators. Efficacy and safety of alirocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1489-99. doi: 10.1056/NEJMoa1501031. Epub 2015 Mar 15. PMID 25773378
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Kastelein JJ, Hovingh GK, Langslet G, Baccara-Dinet MT, Gipe DA, Chaudhari U, Zhao J, Minini P, Farnier M. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 monoclonal antibody alirocumab vs placebo in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Jan-Feb;11(1):195-203.e4. doi: 10.1016/j.jacl.2016.12.004. Epub 2016 Dec 28. PMID 28391886
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 320 centers in 27 countries. Overall, 5144 participants were screened between January 2012 and March 2013, 2801 of whom were screen failures. Screen failures were mainly due to exclusion criteria met. In addition 2 participants received study drug but did not undergo randomization. They were excluded from analysis.
Pre-assignment Details: Randomization was stratified as per diagnosis of heterozygous familial hypercholesterolemia (heFH), prior history of myocardial infarction (MI) or ischemic stroke, intensity of statin treatment and geographic region. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:2 ratio (placebo:alirocumab).
Groups:
- Placebo Q2W: Placebo (for alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable lipid modifying therapy (LMT) for 78 weeks.
- Alirocumab 150 mg Q2W: Alirocumab 150 mg SC injection Q2W added to stable LMT for 78 weeks.
Period: Overall Study
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Started | 788 (Randomized) | 1553 (Randomized)
Treated | 788 | 1550
Completed | 595 | 1113
Not Completed | 193 | 440
Not completed — Randomized but not treated | 0 | 3
Not completed — Adverse Event | 48 | 113
Not completed — Death | 6 | 2
Not completed — Poor compliance to protocol | 38 | 60
Not completed — Physician Decision | 0 | 4
Not completed — Participant moved | 5 | 19
Not completed — Consent withdrawn by participant | 34 | 72
Not completed — Related to study drug administration | 5 | 14
Not completed — Last visit outside protocol visit window | 51 | 143
Not completed — Selection criteria finally not met | 0 | 1
Not completed — Site closure | 0 | 3
Not completed — Potential lost to follow-up | 3 | 0
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo Q2W: Placebo (for alirocumab) SC injection Q2W added to stable LMT for 78 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W | Total
Number analyzed (Participants) | 788 | 1553 | 2341
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.4) | 60.4 (10.4) | 60.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 570 | 884
  Male | 474 | 983 | 1457
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol - [Triglyceride/5]).
  mg/dL | 121.9 (41.4) | 122.7 (42.6) | 122.4 (42.2)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.157 (1.073) | 3.178 (1.102) | 3.171 (1.092)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events (AEs)
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Time Frame: Up to 10 weeks after last study drug administration (maximum of 86 weeks)
Population: Safety population: all randomized participants who received at least one dose or part of a dose of a study drug (treated).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 788 | 1550
percentage of participants
  Any AE | 82.5 | 81.0
  Any Serious AE | 19.5 | 18.7
  Any AE leading to death | 1.3 | 0.5
  Any AE leading to treatment discontinuation | 5.8 | 7.2

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Adjusted least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 0.8 (1.0) | -61.0 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -61.9, 95% CI 2-sided [-64.3 to -59.4] — Alirocumab vs. Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percent change | 0.7 (1.0) | -62.8 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; A hierarchial testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchial testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -63.5, 95% CI 2-sided [-65.9 to -61.2] — Alirocumab vs. Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 1.5 (1.0) | -63.3 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -64.8, 95% CI 2-sided [-67.2 to -62.4] — Alirocumab vs. Placebo

5. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percent change | 1.4 (1.0) | -64.2 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -65.5, 95% CI 2-sided [-67.9 to -63.2] — Alirocumab vs. Placebo

6. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 24 - ITT Analysis
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline measured LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 652 | 1278
percent change | 3.5 (1.1) | -57.8 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -61.3, 95% CI 2-sided [-64.0 to -58.5] — Alirocumab vs. Placebo

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 753 | 1468
percent change | 1.2 (1.0) | -52.8 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -54.0, 95% CI 2-sided [-56.3 to -51.7] — Alirocumab vs. Placebo

8. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo-B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 743 | 1444
percent change | 1.2 (0.9) | -54.3 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -55.5, 95% CI 2-sided [-57.7 to -53.2] — Alirocumab vs. Placebo

9. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 0.7 (0.9) | -51.6 (0.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -52.3, 95% CI 2-sided [-54.4 to -50.2] — Alirocumab vs. Placebo

10. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percent change | 0.6 (0.9) | -53.1 (0.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -53.7, 95% CI 2-sided [-55.7 to -51.6] — Alirocumab vs. Placebo

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | -0.3 (0.7) | -37.8 (0.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -37.5, 95% CI 2-sided [-39.1 to -35.9] — Alirocumab vs. Placebo

12. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 753 | 1468
percent change | 0.5 (0.9) | -55.5 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -56.0, 95% CI 2-sided [-58.3 to -53.7] — Alirocumab vs. Placebo

13. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 12
Time Frame: From Baseline to Week 52
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 0.9 (0.8) | -53.7 (0.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -54.6, 95% CI 2-sided [-56.6 to -52.6] — Alirocumab vs. Placebo

14. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 12
Time Frame: From Baseline to Week 52
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 0.2 (0.6) | -38.8 (0.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -39.0, 95% CI 2-sided [-40.4 to -37.5] — Alirocumab vs. Placebo

15. Secondary Outcome: Percentage of Very High Cardiovascular (CV) Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Very high CV risk: Heterozygous Familial Hypercholesterolemia (heFH) participants with coronary heart disease (CHD) or CHD risk equivalents or non- Familial Hypercholesterolemia (FH). High CV risk: heFH participants without CHD or CHD risk equivalents. CHD risk equivalent: peripheral arterial disease, ischemic stroke, moderate chronic kidney disease (estimated glomerular filtration rate, 30 to <60 ml/minute/1.73 m^2 of body-surface area), or diabetes mellitus plus 2 or more additional risk factors (hypertension; ankle-brachial index of ≤0.90; microalbuminuria, macroalbuminuria, or a urinary dipstick result of >2+ protein; preproliferative or proliferative retinopathy or laser treatment for retinopathy; or family history of premature CHD). Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percentage of participants | 8.5 | 80.7
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 71.5, 95% CI 2-sided [51.6 to 99.1] — Alirocumab vs. Placebo

16. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were from multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percentage of participants | 8.5 | 82.8
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 93.4, 95% CI 2-sided [66.1 to 132.0] — Alirocumab vs. Placebo

17. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percentage of participants | 8.0 | 79.3
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 74.6, 95% CI 2-sided [53.3 to 104.4] — Alirocumab vs. Placebo

18. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including available post-baseline data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percentage of participants | 8.0 | 81.2
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 97.3, 95% CI 2-sided [68.2 to 138.9] — Alirocumab vs. Placebo

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | -3.7 (1.0) | -29.3 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -25.6, 95% CI 2-sided [-28.1 to -23.1] — Alirocumab vs. Placebo

20. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | -0.6 (0.5) | 4.0 (0.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 4.6, 95% CI 2-sided [3.3 to 5.9] — Alirocumab vs. Placebo

21. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 1.8 (1.2) | -15.6 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -17.3, 95% CI 2-sided [-20.1 to -14.6] — Alirocumab vs. Placebo

22. Secondary Outcome: Percent Change From Baseline in Apo A1 at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A1 value on- or off-treatment (Apo A1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 753 | 1468
percent change | 1.2 (0.6) | 4.0 (0.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 2.9, 95% CI 2-sided [1.6 to 4.2] — Alirocumab vs. Placebo

23. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | -3.1 (1.0) | -28.2 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -25.1, 95% CI 2-sided [-27.4 to -22.7] — Alirocumab vs. Placebo

24. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 12
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 0.2 (0.5) | 5.8 (0.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 5.6, 95% CI 2-sided [4.3 to 6.8] — Alirocumab vs. Placebo

25. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 23
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 1.2 (1.1) | -16.7 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -17.9, 95% CI 2-sided [-20.5 to -15.3] — Alirocumab vs. Placebo

26. Secondary Outcome: Percent Change From Baseline in Apo A1 at Week 12 - ITT Analysis
Description: as for outcome 12
Time Frame: From Baseline to Week 52
Population: Apo A1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 753 | 1468
percent change | 0.6 (0.5) | 4.6 (0.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 4.0, 95% CI 2-sided [2.8 to 5.2] — Alirocumab vs. Placebo

27. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 4.4 (1.2) | -56.8 (0.8)

28. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percent change | 4.6 (1.1) | -59.9 (0.8)

29. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM model including all available post-baseline data from Week 4 to Week 78 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 78
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 780 | 1530
percent change | 3.6 (1.3) | -52.4 (0.9)

30. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 78 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 78
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 777 | 1523
percent change | 3.9 (1.2) | -58.0 (0.9)

31. Other Pre Specified Outcome: Percentage of Participants Who Experienced Cardiovascular (CV) Events
Description: CV events included coronary heart disease (CHD) death; non-fatal myocardial infarction (MI); fatal and non-fatal ischemic stroke; unstable angina requiring hospitalization; congestive heart failure (CHF) requiring hospitalization; ischemia-driven coronary revascularization procedure. Reported events are CV events as confirmed by an independent Clinical Events Committee (CEC) that occurred during the treatment emergent period ( i.e. from first dose up to the last dose of study drug + 70 days).
Time Frame: Up to 10 weeks after last study drug administration (maximum of 86 weeks)
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 788 | 1550
percentage of participants | 5.1 | 4.6

32. Post Hoc Outcome: Percentage of Participants Who Experienced Major Adverse CV Events
Description: Major adverse CV events were defined as all adverse CV events except Congestive heart failure (CHF) requiring hospitalization; and ischemia-driven coronary revascularization procedure.
Time Frame: Up to 10 weeks after last study drug administration (maximum of 86 weeks)
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 788 | 1550
percentage of participants | 3.3 | 1.7

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 86 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 154/788 | 290/1550
Other Adverse Events (participants affected / at risk) | 366/788 | 707/1550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=788) | Alirocumab 150 mg Q2W (N=1550)
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 5
Pneumonia (Infections and infestations) | 7 | 6
Cellulitis (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 1 | 5
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 8
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleomorphic liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Thyrotoxic crisis (Endocrine disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Lipomatosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2
Major depression (Psychiatric disorders) | 1 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 6 | 11
Hypoaesthesia (Nervous system disorders) | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 7
Presyncope (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 5
Migraine (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 2
Loss of consciousness (Nervous system disorders) | 0 | 3
Carotid arteriosclerosis (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 3
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Nerve root compression (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 1
Demyelination (Nervous system disorders) | 0 | 1
Frontotemporal dementia (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Miller Fisher syndrome (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Endocrine ophthalmopathy (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1
Blepharochalasis (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 9 | 29
Angina pectoris (Cardiac disorders) | 6 | 9
Atrial fibrillation (Cardiac disorders) | 7 | 9
Cardiac failure (Cardiac disorders) | 3 | 4
Coronary artery disease (Cardiac disorders) | 3 | 10
Acute myocardial infarction (Cardiac disorders) | 11 | 9
Bradycardia (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 2 | 3
Cardiac failure chronic (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 4
Myocardial infarction (Cardiac disorders) | 4 | 4
Ventricular tachycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 3
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 6 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 4
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 3 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 8
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Cystitis interstitial (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 13
Chest pain (General disorders) | 1 | 0
Coronary artery restenosis (General disorders) | 1 | 1
Device failure (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 4 | 1
Peripheral artery restenosis (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=788) | Alirocumab 150 mg Q2W (N=1550)
Nasopharyngitis (Infections and infestations) | 103 | 209
Upper respiratory tract infection (Infections and infestations) | 68 | 114
Urinary tract infection (Infections and infestations) | 54 | 87
Influenza (Infections and infestations) | 43 | 88
Bronchitis (Infections and infestations) | 40 | 83
Headache (Nervous system disorders) | 44 | 76
Diarrhoea (Gastrointestinal disorders) | 45 | 89
Back pain (Musculoskeletal and connective tissue disorders) | 52 | 84
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 84
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 | 80
Injection site reaction (General disorders) | 33 | 91

LIMITATIONS AND CAVEATS:
Manual reclassification was done by the Sponsor for the "other reasons" of non-completion of study as specified in the electronic case report (eCRF) form.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.